CLINICAL TRIAL: NCT05304065
Title: Youth Partners in Care for Suicide Prevention
Brief Title: Safe Treatment for Emergency Presentation for Suicidal Ideation and Behavior in Youth
Acronym: SAFE STEPS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Duke University (Other); Brown University (Other); University of Utah (Other); Olive View-UCLA Education & Research Institute (Other); RAND (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Joan Asarnow, Professor of Psychiatry & Biboehavioral Sciences, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SP-2020C3-21078
Record Dates: First submitted 2022-03-11; First posted 2022-03-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Suicide; Suicidal; Self-Harm
Keywords: self-harm
MeSH Terms: conditions — Suicide; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: It is not possible to mask intervention condition from participants. Care providers in the ED will be masked to randomized condition. Outcomes assessors will be masked to randomized condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAFETY-Acute within Usual ED Care (Active Comparator): The SAFETY-Acute (A) approach to safety planning and stabilization will be integrated within usual ED Care. SAFETY-A was formerly called the Family Intervention for Suicide Prevention, FISP.
  Interventions: Behavioral: SAFETY-A within usual ED Care
- Combined (Active Comparator): The combined treatment arm includes both 1) SAFETY-A integrated within usual ED Care, and 2) therapeutic follow-up contacts using the Coping Long Term with Active Suicidality Program (CLASP) model.
  Interventions: Behavioral: Combined SAFETY-A within usual ED Care + CLASP Therapeutic Follow-Up Contacts

INTERVENTIONS:
Behavioral: SAFETY-A within usual ED Care — SAFETY-A is a single session collaborative, strengths-based, developmentally nuanced, cognitive-behavioral intervention (CBT) to increase safety and mental health treatment initiation. The therapist works with the youth and family (or significant other, SO) separately and together to build hope and reasons for living, develop a personal safety plan, increase protective supports; and increase motivation for and linkage to treatment.
  Other Names: Family Intervention for Suicide Prevention (FISP)
  Arms: SAFETY-Acute within Usual ED Care
Behavioral: Combined SAFETY-A within usual ED Care + CLASP Therapeutic Follow-Up Contacts — COMB, includes SAFETY-A within usual ED care plus CLASP therapeutic and caring follow-up contacts designed to strengthen safety and treatment initiation and engagement. Core functions of CLASP include: building hope/reducing hopelessness; enhancing social/family support; strengthening problem-solving; and increasing treatment initiation and engagement.
  Arms: Combined

SUMMARY:
This randomized comparative effectiveness trial will compare two evidence-based approaches to emergency care for youth ages 13-24 who present to the Emergency Department (ED) with suicidal ideation or behavior. Outcomes will be monitored at baseline and at 3, 6 & 12 month follow-up assessments.

DETAILED DESCRIPTION:
Rationale and Importance of Study:

Suicide is currently the second leading cause of death for U.S. youth ages 13-24, responsible for more deaths than any major illness. Youth with serious suicidal behavior or thoughts often present to the nation's Emergency Departments (EDs), particularly youth who make potentially deadly suicide attempts. Evidence is limited regarding optimal interventions for reducing the risk of fatal and nonfatal suicide attempts in these youth, and tested interventions include multiple components. One dimension along which these interventions vary is timing. Some interventions are delivered in the ED, others focus on aftercare, and others combine ED and aftercare interventions. Current evidence supports effectiveness of some interventions for reducing later suicide attempts and improving the likelihood that youth will receive mental health treatment after leaving the ED. However, evidence gaps exist regarding: 1) whether it is sufficient to focus on providing an evidence-based intervention in the ED, or whether a post-ED aftercare intervention is needed to improve youth outcomes; and 2) for which patient subgroups a combined ED and aftercare treatment may be indicated. Answering these questions is vital for guiding resource allocation, as ED care emphasizes care in the ED with limited resources for aftercare.

Study Aims:

The study addresses this evidence gap by comparing two evidence-based interventions for reducing suicide attempts and improving outcomes for youth presenting to EDs with suicidal episodes: 1) Safety-Acute(A) integrated within ED care, a crisis therapy/safety planning intervention in the ED focused on enhancing safety (previously called Family Intervention for Suicide Prevention, FISP); and 2) SAFETY-A/ED care plus the Coping Long-term with Active Suicide Program (CLASP), comprised of brief therapeutic follow-up contacts after discharge from the ED/hospital. Evidence supports benefits of both interventions individually. SAFETY-A/FISP is listed in the National Register of Evidence-Based Practices, and CLASP is being implemented in some Veterans Administration Hospitals. The first aim is to evaluate whether SAFETY-A/ED Care combined with CLASP aftercare is superior to SAFETY- A/ED Care alone for reducing the risk of suicide attempts and increasing initiation of follow-up mental health treatment. Second, the investigators examine heterogeneity of treatment effects among subgroups, hypothesizing that in this large diverse sample the strongest benefits of the combined SAFETY-A/ED Care plus CLASP intervention will be seen in youth who are from ethnic or racial minority groups, socioeconomically disadvantaged, and from rural communities. Third, the investigators aim to increase the value and relevance of the study by engaging patients, parents, family members, providers, and health and mental healthcare system stakeholders in project leadership and activities throughout the study and implement a partnered dissemination plan to enhance the potential for study findings to inform clinical practice and health care delivery.

Study Description:

The patient population includes 1,600 youth ages 13-24 presenting to EDs with suicidal ideation or behavior in 4 communities across the country selected to include a diverse population (racial, ethnic, rural vs urban, public vs private insurance): California/Los Angeles; North Carolina; Rhode Island; Utah. Youth are randomly assigned to: 1) SAFETY-A/ED Care; or 2) SAFETY-A/ED Care plus CLASP. Assessments are conducted at the start of the study and at 3, 6, and 12-month follow-ups. Primary outcomes are suicide attempts and mental health treatment initiation. Secondary outcomes are overall self-harm (including suicide attempts and non-suicidal self-harm) and treatment engagement/dose. Exploratory outcomes are: severity of youth suicidality; youth functioning and quality of life; and improvement on three problems prioritized by the youth and parent or significant other as "top problems." The investigators also examine change in identified protective and risk factors (e.g. connectedness, hopelessness, and perceived barriers to treatment). The investigators partner with diverse stakeholders, develop a Stakeholder Council, and include stakeholder partners in project leadership and activities with the goals of promoting 2-way knowledge exchange and enhancing the value of the study for improving patient care and outcomes.

Significance:

Study results will clarify whether the additional resources needed to provide brief therapeutic follow-up calls after an ED intervention leads to improved outcomes, and which patient subgroups are most likely to benefit from a treatment approach that provides therapeutic contact both during the ED visit and after discharge from the ED. This information can guide decision makers regarding how to best develop services and service systems to improve patient outcomes and achieve national suicide prevention goals, including for diverse groups to improve equity.

ELIGIBILITY:
Inclusion Criteria:

* age 13-24;
* past-week suicidal behavior or ideation with plan or intent

Exclusion Criteria:

* symptoms or illness that precludes informed consent or engagement in study procedures (e.g., active psychosis; drug dependence, no locator information);
* youth not fluent in English
* parent not fluent in English or Spanish.

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1600 (Estimated)
Dates: Start 2022-10-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Suicide Attempts: Primary Clinical Outcome | Through 12 months of follow-up
  suicide attempts fatal, nonfatal, and interrupted
Mental Health Treatment Initiation: Primary Service Use Outcome | Observed through 12 months of follow-up, primary end point 6-month follow-up
  initiation of mental health treatment after discharge from ED/hospital

SECONDARY OUTCOMES:
Self-Harm: Secondary Clinical Outcome | Through 12 months of follow-up
  Any self-harm including suicidal, nonsuicidal, and ambiguous self-harm
Treatment engagement: Secondary Service Use Outcome | Through 12 months of follow-up
  Treatment dose received

OTHER OUTCOMES:
Ordinal suicidality scale: Clinical | Through 12 months of follow-up
  Ranges from nonsuicidal through ideation, behavior, attempts, and deaths
Quality of life and functioning: Clinical | Change from baseline through 12 months of follow-up
  PROMIS Global Health Questionnaire , 0-100

CONTACTS AND LOCATIONS:
Overall Officials: Joan R Asarnow, PhD, Principal Investigator — University of California, Los Angeles; David Goldston, PhD, Principal Investigator — Duke University
Locations (5):
- United States (5):
  - Ronald Reagan Medical Center, Los Angeles, California
  - Olive View UCLA Education and Research Center, Sylmar, California
  - Duke University, Durham, North Carolina
  - Brown University, Providence, Rhode Island
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Decision will be made with PCORI, project investigators, and stakeholders regarding any data sharing. Given relative rarity of suicide attempts it is critical that participant confidentiality be maintained and steps be taken to protect against the possible of unintended loss of anonymity due to focus on rare outcome.
Supporting Information: Study Protocol
Time Frame: A limited data set may be available after all data are complete, analyzed, and published. Time frame and plan will be developed by investigators in collaboration with stakeholders and funding agency (PCORI).
Access Criteria: Decision will be made with PCORI, project investigators, and stakeholders regarding any data access. Given rarity of suicide attempts it is critical that participant confidentiality be maintained and steps be taken to protect against the possibility of unintended loss of anonymity due to focus on rare outcomes.

REFERENCES:
- See also: Study description on PCORI site — http://www.pcori.org/research-results/2021/youth-partners-care-suicide-prevention-ypic-sp